CLINICAL TRIAL: NCT05535998
Title: TACE-HAIC Combined With Targeted Therapy and Immunotherapy Versus TACE Alone for Hepatocellular Carcinoma With Portal Vein Tumor Thrombus: A Propensity Score Matching Study
Brief Title: TACE-HAIC Combined With TKIs and Immunotherapy Versus TACE Alone for Hepatocellular Carcinoma With PVTT
Status: Completed | Type: Observational
Sponsor: Yunfei Yuan (Other)
Responsible Party: Sponsor-Investigator, Yunfei Yuan, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Other Study IDs: B2022-312-01
Record Dates: First submitted 2022-09-08; First posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC; TACE-HAIC; TACE; TKIs; PD-1 Inhibitors
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Immune Checkpoint Inhibitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Combined therapy group (TACE-HAIC combined with TKIs and PD-1 inhibitors): Patients recieve combined with TKIs and PD-1 inhibitors
  Interventions: Procedure: TACE-HAIC; Drug: Targeted therapy; Drug: PD-1 inhibitors
- TACE alone group: TACE alone
  Interventions: Procedure: TACE

INTERVENTIONS:
Procedure: TACE-HAIC — The TACE-HAIC which was performed using 30 mg/m2 of epirubicin mixed with 2-5 mL lipiodol, followed by pure lipiodol. Then, a catheter was placed and fixed in the tumor feeding artery for the FOLFOX-based chemotherapy infusion at the following dosage: 85 mg/m2 of oxaliplatin infusion for 2 hours; leucovorin, 400 mg/m2 infusion for 2 hours; 400 mg/m2 of 5-FU bolus; and 2400 mg/m2 of continuous 5-FU infusion for 46 hours or 1200mg/m2 of continuous 5-FU infusion for 23 hours, respectively. Repeated TACE-HAIC was performed at intervals of 3-4 weeks.
  Groups: Combined therapy group (TACE-HAIC combined with TKIs and PD-1 inhibitors)
Procedure: TACE — TACE was performed using 30 mg/m2 of epirubicin, 200 mg/m2 of carboplatin, and 4mg/m2 of MMC, mixed with 2-5 mL lipiodol. Up to 20 mL of additional pure lipiodol were injected into the tumor-feeding artery until stasis of blood flow was observed in the target artery. Repeated TACE was performed at intervals of 3-4 weeks.
  Groups: TACE alone group
Drug: Targeted therapy — The TKI therapy used in this study were lenvatinib (12 mg/d for bodyweight ⩾ 60 kg or 8 mg/d for bodyweight <60 kg), sorafenib (400 mg twice a day) or apatinib (250-500 mg orally once daily). Administration of lenvatinib, apatinib or sorafenib was started on the first post-TACE day, and continually administered until disease progression developed or serious treatment-related toxicity occurred.
  Groups: Combined therapy group (TACE-HAIC combined with TKIs and PD-1 inhibitors)
Drug: PD-1 inhibitors — PD-1 inhibitors were intravenously administered on the first post-TACE day as follows: camrelizumab 200 mg or sintilimab 200 mg or toripalimab 240 mg or tislelizumab 200 mg, every 3-4 weeks.
  Groups: Combined therapy group (TACE-HAIC combined with TKIs and PD-1 inhibitors)

SUMMARY:
Hepatocellular carcinoma (HCC) is characterized with vascular invasion, particularly of the portal vein, resulting in portal vein tumor thrombus (PVTT) in 10%-40% of HCC patients at the time of HCC diagnosis. The prognosis of these patients is extremely poor.Treatment efficacy and safety using a combined therapy (TACE-HAIC combined with TKIs and PD-1 inhibitors) were compared with TACE alone in treatment of HCC patients with PVTT.

ELIGIBILITY:
Inclusion Criteria:

* (a) HCC patients with PVTT (Vp1-4) treated by TACE, or the combination therapy (TACE-HAIC combined with TKIs or an PD-1 inhibitors) as initial treatment; (b) age between 18 and 75 years; (c) Child-Pugh A or B liver function; (d) Eastern Cooperative Oncology Group (ECOG) performance status 0-1; (e) adequate hematologic blood counts (white blood cell count >3ⅹ109/L, absolute neutrophil count >1.5ⅹ109/L, platelet count >10ⅹ109/L, hemoglobin concentration >85 g/L); (f) no extrahepatic metastasis.

Exclusion Criteria:

* (a) severe underlying cardiac, pulmonary, or renal diseases; (b) history of a second primary malignant tumor; (c) incomplete medical data; (d) loss to follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We reviewed data of 743 patients diagnosed as HCC patients with PVTT at Sun Yat-Sen University Cancer Center. 604 patients received TACE, and 139 patients received combination therapy.
Sampling Method: Non-Probability Sample
Enrollment: 743 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Tumor Response | 24 months
  The tumor responses were evaluated by measuring the longest diameter of target lesions according to response evaluation criteria in solid tumors (RECIST) version 1.1
Overall survival | 24 months
  Overall survival (OS) was measured from the initiation of transarterial therapy to the date of death or the last follow-up.
Progression-free survival | 24 months
  Progression-free survival (PFS) was measured from the initiation of transarterial therapy to the time of progression or recurrence or last follow-up.

SECONDARY OUTCOMES:
Conversion rate | 24 rates
  Rate of patients underwent hepatic surgery after careful evaluation when an estimated residual liver volume >30-40% could be remained after R0 surgery by 2 experienced surgeons

CONTACTS AND LOCATIONS:
Overall Officials: Yunfei Yuan, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No